CLINICAL TRIAL: NCT06715865
Title: Clinical Study on Thymus-Kidney Transplantation From Neonatal Donors for the Induction of Immune Tolerance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2024-248-B
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thymus Transplantation Group (Experimental)
  Interventions: Procedure: Thymus Transplantation

INTERVENTIONS:
Procedure: Thymus Transplantation — Thymus Transplantation

SUMMARY:
Thymus transplantation for the induction of immune tolerance in kidney transplantation: This study aims to understand how thymus transplantation can induce immune tolerance in recipients of allogeneic kidney transplants to achieve the discontinuation of immunosuppressive therapy. It will evaluate the safety of thymus transplantation, explore the functional output of thymus tissue, investigate the optimal timing for withdrawal of immunosuppressants, and identify key indicators for the reconstruction of immune suppression capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Recipients of both thymus and kidney transplants from the same donor.
2. Age between 18 and 65 years.
3. Non-solid organ combination transplant recipients (including heart-kidney or liver-kidney transplants, except thymus).
4. ABO blood type compatibility with the donor.
5. Negative donor-specific antibody (DSA).
6. Negative lymphocyte crossmatch (CDC).
7. Normal cardiac function (confirmed through ECG and echocardiograms).
8. Normal liver function.
9. Bodyweight between 40-100 kg (inclusive).
10. Evidence of prior epstein-barr virus (EBV) infection with positive EBV-specific immunoglobulin G (IgG) and negative immunoglobulin M (IgM).
11. Signed informed consent form.
12. Ability to adhere to regular follow-ups.
13. Normal hematopoietic function.

Exclusion Criteria:

1. Clinically significant genital or urinary tract dysfunction.
2. Underlying kidney diseases with a high risk of recurrence in the transplanted kidney, including:

   * a. Focal segmental glomerulosclerosis (FSGS).
   * b. Type I or II membranoproliferative glomerulonephritis.
   * c. Hemolytic uremic syndrome/thrombotic thrombocytopenic purpura (HUS/TTP).
3. Any genetic mutation-associated diseases.
4. Presence of infectious diseases:
5. Strongly positive panel reactive antibodies (PRA).
6. History of receiving blood transfusion therapy.
7. Any other conditions that, in the investigator's opinion, are incompatible with participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Duration of immunosuppressive therapy after surgery | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China